CLINICAL TRIAL: NCT00390416
Title: A Phase II Study of Docetaxel, Cisplatin, and Fluorouracil (Modified DCF) With Bevacizumab in Patients With Unresectable or Metastatic Gastroesophageal Adenocarcinoma
Brief Title: Study of Docetaxel, Cisplatin, and Fluorouracil (Modified DCF) With Bevacizumab in Patients With Unresectable or Metastatic Gastroesophageal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sanofi (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-096; NCT00403468 (obsolete NCT alias)
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
Keywords: Metastatic; Gastroesophageal; Docetaxel; Cisplatin; Fluorouracil; Bevacizumab; Metastatic Gastroesophageal Adenocarcinoma; 06-096
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Cisplatin; Fluorouracil; Bevacizumab; Leucovorin

ARMS (1):
- Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin (Experimental): Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
  Interventions: Drug: Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin — Bevacizumab 10mg/kg day 1 IV over 30 minutes Docetaxel 40mg/m2 day 1 IV over 1 hour Leucovorin 400mg/m2 day 1 IV over 30 minutes Fluorouracil 400mg/m2 IVP day 1 Fluorouracil 1000mg/m2 IVCI x 48 hours Cisplatin 40mg/m2 day 3 IV over 30 minutes

SUMMARY:
This study is being done to find out what effects a drug named/called bevacizumab has on patients and patients' tumors when given together with standard chemotherapy drugs. Making new blood vessels seems to be important for many tumors to grow. Bevacizumab is a new type of treatment for cancer that blocks the growth of new tumor blood vessels. In this study, the researchers will combine bevacizumab with chemotherapy drugs that are standard for the patient's disease and include cisplatin, docetaxel, fluorouracil, and leucovorin. The way the original combination of cisplatin, docetaxel, and fluorouracil was given caused many side effects including gastrointestinal symptoms, weakness, and a drop in the blood count of infection fighting cells. For this study, the researchers have modified this combination to give lower doses of the medicines more often, to reduce side effects from the chemotherapy. Patients will receive bevacizumab with this modified combination of docetaxel, cisplatin, and fluorouracil. This study is called a phase II study. In this study, everyone will have similar tumors and receive the same treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or unresectable gastric or esophageal adenocarcinoma, including GEJ adenocarcinoma which will be classified according to Siewert's classification type I, II, or III.
* Histological documentation of local recurrence or metastasis is strongly encouraged, unless the risk of such a procedure outweighs the potential benefit of confirming the metastatic disease.
* If no histologic confirmation, then the metastases or recurrence will require documentation by a 2nd radiographic procedure (i.e. positron emission tomography [PET] scan or magnetic resonance imaging [MRI] in addition to the computed tomography [CT] scan). If the imaging procedure does not confirm recurrent or metastatic disease, biopsy confirmation will be required.
* Patients must have disease that can be evaluated radiographically. This may be measurable disease or non-measurable disease. Measurable disease is defined as that which can be measured in at least one dimension as > or = 20 mm with conventional techniques, or > or = 10 mm by high resolution imaging. Disease that is identified on radiology studies, but does not meet the criteria for measurable disease, is considered non-measurable - see section 12.1.1 of protocol for further details.
* No prior chemotherapy for metastatic or unresectable disease. Patients may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if more than 6 months have elapsed between the end of adjuvant therapy and registration. Patients may not have received prior docetaxel or cisplatin, or bevacizumab or any other novel biologic anti-angiogenic agent.
* Age 18 years or older.
* Karnofsky performance status > or = 70% (ECOG performance status 0-1).
* Peripheral neuropathy < or = grade 1
* Hematologic (minimal values):

  * White blood cell count > or = 3000/mm3
  * Absolute neutrophil count > or = 1500 cells/mm3
  * Hemoglobin > or = 9.0 g/dl
  * Platelet count > or = 100,000/mm3
* Hepatic (minimal values):

  * Total bilirubin < or = to upper limit of normal (ULN)
  * AST and ALT and alkaline phosphatase must be within the eligible range. In determining eligibility, the more abnormal of the two values (AST or ALT) should be used. AST and ALT and alkaline phosphatase should be no more than 1-1.5 times the upper limit of normal.
* Kidney function (minimal values):

  * Serum creatinine < or = 1.5 mg/dl
  * Urinalysis < 2+ proteinuria; urine protein (mg/dl)/urine creatinine (mg/dl) ratio (Up/c) < 1.0
* The patient has a PT (INR) < or = 1.5 and a PTT < or = 3 seconds above the upper limits of normal if the patient is not on anticoagulation therapy. If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:

  1. The patient must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW heparin.
  2. The patient must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices).
* Women of childbearing potential must have a negative pregnancy test. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Ability to understand informed consent and signing of written informed consent document prior to initiation of protocol therapy.

Exclusion Criteria:

* Patients who have received previous chemotherapy for the treatment of metastatic or unresectable gastric, GEJ, or esophageal adenocarcinoma are ineligible. Patients who have received previous pre- or post-operative chemotherapy or chemoradiation are ineligible if therapy was completed less than 6 months prior to study registration. Patients must have recovered from adverse events from any previous therapy.
* Patients who have received previous bevacizumab, docetaxel, or cisplatin.
* Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
* Patients with brain or central nervous system metastases, including leptomeningeal disease.
* Minor surgical procedure such as fine needle aspiration, core biopsy, laparoscopy, or mediport placement within 7 days prior to initiating treatment.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0
* Anticipation of need for major surgical procedure during the course of the study.
* Pregnant (positive pregnancy test) or breast feeding.
* Urine protein:creatinine (Up/c) ratio > or = 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to the initiation of treatment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Blood pressure > 150/100 mmHg
* Significant cardiac disease defined as:

  * Unstable angina
  * New York Heart Association (NYHA) grade II or greater
  * Congestive heart failure
  * History of myocardial infarction within 6 months
* Evidence of bleeding diathesis or coagulopathy.
* History of a stroke or cerebrovascular accident (CVA) within 6 months.
* Clinically significant peripheral vascular disease.
* Clinically significant hearing loss or ringing in the ears.
* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80.
* Inability to comply with study and/or follow-up procedures.
* Patients with any other medical condition or reason, in the investigator's opinion, that makes the patient unstable to participate in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ilson, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
Started | 48
Completed | 44
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Not treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival
Description: as measured from the start of the treatment to the date of either documentation of disease progression or death. As we have previously, we will define progression of disease as per RECIST criteria. As per RECIST criteria, any evidence of progression in non-measurable lesions, measurable lesions, or the development of new lesions, would qualify as disease progression .RECIST criteria as defined by CTEP (http://ctep.info.nih.gov/Policies).
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
Number analyzed (Participants) | 39
percentage of participants | 79 [63 to 88]

2. Secondary Outcome: Patients With Measurable Disease the Confirmed Response Rate
Time Frame: up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
Number analyzed (Participants) | 39
percentage of participants
  Confirmed Response Rate | 67 [50 to 81]
  Response Rate (proximal/GEJ tumors) | 85 [62 to 97]

3. Primary Outcome: 1-year Survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
Number analyzed (Participants) | 39
months
  Progression Free Survival | 12 [8.8 to 1832]
  Overall Survival | 16.8 [12.1 to 26.1]

ADVERSE EVENTS:
Arm/Group | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin
Serious Adverse Events (participants affected / at risk) | 27/48
Other Adverse Events (participants affected / at risk) | 44/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin (N=48)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection, other (Infections and infestations) | 3 (4)
White blood cell decreased (Investigations) | 1 (1)
Mucositis-Oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Neutrophil count decreased (Investigations) | 8 (9)
Rectal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Chest pain-cardiac (Cardiac disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Platelet count decrease (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Cisplatin, Fluorouracil, Bevacizumab, Leucovorin (N=48)
Alanine aminotransferase increase (Investigations) | 4 (6)
Aspartate aminotransferase increase (Investigations) | 5 (9)
Allergic reaction (Immune system disorders) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 5 (7)
Creatinine increased (Investigations) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 8 (15)
Diarrhea (Gastrointestinal disorders) | 13 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 4 (6)
Fatigue (General disorders) | 28 (104)
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 3 (18)
Anemia (Blood and lymphatic system disorders) | 26 (241)
White blood cell decreased (Investigations) | 36 (197)
Lymphocyte count decreased (Investigations) | 26 (115)
Hypomagnesemia (Metabolism and nutrition disorders) | 20 (112)
Mucositis-Oral (Gastrointestinal disorders) | 20 (37)
Nausea (Gastrointestinal disorders) | 12 (24)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (54)
Neutrophil count decreased (Investigations) | 34 (127)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 30 (119)
Platelet count decreased (Investigations) | 11 (58)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (6)
Dysgeusia (Nervous system disorders) | 4 (4)
Thrombosis/thrombus/embolism (Vascular disorders) | 19 (21)
Tinnitus (Ear and labyrinth disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 5 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes